CLINICAL TRIAL: NCT02860247
Title: Rapid Detection of Bacterial Resistance by MALDI-TOF MS and Antibiotic Savings
Acronym: MALDI-TRAc
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2016/300
Record Dates: First submitted 2016-08-01; First posted 2016-08-09 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Sepsis With Escherichia Coli
Keywords: antibiotic; MALDI-TOF MS; susceptibility testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims at determining within a short time (<3h) the susceptibility to clinical isolates of E. coli to the major antibiotics directly from positive blood cultures.

DETAILED DESCRIPTION:
The resistance to antibiotic is a concern for the great majority of pathogenic bacteria. The proportion of antibiotic-resistant bacteria is particularly high in hospital settings. The accumulation of resistance mechanisms can lead to multidrug resistance, therapeutic impasses and a subsequent higher mortality of infected patients. The use of antibiotics in humans and animals creates a selection pressure that favors the dissemination of antibiotic resistant strains. It's necessary to optimize antibiotic consumption to limit the spread of these bacteria. It requires both the fast bacterial identification and the fast determination of their resistance profile in order to use narrower-spectrum compounds.

Usually antibiotic susceptibility testing usually takes 18-24 hours. Mass Spectrometry type Matrix-Assisted Laser Desorption Ionization Time-Of-Flight (MALDI-TOF MS) has become a valuable tool in clinical laboratories for pathogen identification. Preliminary data showed that susceptible and resistant bacteria can be differentiated within 1 or 2 hours with a new technology called 'MS-ASTRA' based on a lower global peak intensity in the presence of the antibiotic of interest (at a concentration corresponding to the susceptibility breakpoint defined by the EUCAST) than in its absence. The objective of this study is to evaluate the performances of this new MALDI-TOF MS method on a panel of wild-type and resistant clinical isolates.

This study aims to determine the resistance of Escherichia coli isolates to cefotaxime, piperacillin-tazobactam, amoxicillin and to implement the method to positive blood cultures. Minimal Inhibitory Concentrations will be determined the standard agar dilution method.

Results and full analyze are deliverable within 2 years. The data obtained with the MS-ASTRA technique will be compared with the resistance status of the clinical isolates. The shortest incubation time (1 or 2 hours) that gives the more accurate result will be evaluate.The antibiotic savings that the implementation of this new method could have allowed will be evaluate.

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized in the hospital of Besançon, with a sepsis with E. coli.

Exclusion Criteria:

* Patients without sepsis with E. coli

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients hospitalized in the hospital of Besançon, with a sepsis with E. coli.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Comparison of antibiotic resistance | Immediate
  assessed by MALDI-TOF MS with that of the reference method (E-test)

SECONDARY OUTCOMES:
Antibiotic savings that could have occurred if the MALDI-TOF MS method was implemented | Immediate
  comparison between the antibiotherapy received by the infected patients (during the first 48 hours) and the adapted treatment which would have been set up from the premature detection of the resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Marlène Sauget, Principal Investigator — CHU Besançon

IPD SHARING:
Plan to Share IPD: No